CLINICAL TRIAL: NCT00163540
Title: Open-Label, Follow-up, Phase IV Clinical Study to Evaluate the Immunogenicity and Safety of a Third Vaccination With FSME-IMMUN 0.5 mL in Subjects Previously Vaccinated Using a Rapid Immunization Schedule (Follow-up to Study 225)
Brief Title: Immunogenicity and Safety Study of a Third Vaccination With FSME-IMMUN 0.5 mL in Subjects Previously Vaccinated According to a Rapid Immunization Schedule (Follow-up to Study 225)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 690501
Record Dates: First submitted 2005-09-08; First posted 2005-09-14 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
Keywords: tick-borne encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: Formaldehyde inactivated, sucrose gradient purified TBE virus antigen, strain Neudörfl

SUMMARY:
The objective of this study is to investigate the immunogenicity and safety of a third vaccination with FSME-IMMUN 0.5 ml given approximately 12 months after the second vaccination in Study 225. In Study 225, two vaccinations were given using a rapid immunization schedule 12 ± 2 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who:
* received 2 vaccinations with FSME-IMMUN 0.5 ml during Study 225
* understand the nature of the study, agree to its provisions and provide written informed consent
* are clinically healthy (i.e. the physician would have no reservation vaccinating with FSME-IMMUN 0.5 ml outside the scope of the clinical trial)
* have a negative pregnancy test result at the first medical examination (if female and capable of bearing children)
* agree to employ adequate birth control measures for the duration of the study (if female and capable of bearing children)
* agree to keep a Subject Diary

Exclusion Criteria:

Subjects who:

* have already been administered a third TBE vaccination elsewhere since receiving two vaccinations in Study 225
* have a history of infection with, or vaccination against, other flaviviruses since participation in Study 225 (e.g. yellow fever, dengue fever, japanese B encephalitis)
* have had an allergic reaction to one of the components of the vaccine since participation in Study 225
* suffer from a disease (e.g. autoimmune disease, immunodeficiency) or are undergoing a form of treatment (e.g., systemic corticosteroids) that can be expected to influence immunological functions
* have a known or suspected problem with drug or alcohol abuse (>4 liters wine/week or equivalent doses of other alcoholic beverages)
* have donated blood or plasma within 30 days of study entry
* have received a blood transfusion or immunoglobulins within 30 days of study entry
* are known to be HIV positive (an HIV test is not required specifically for this study)
* are simultaneously participating in another clinical trial including administration of an investigational product
* have participated in any other clinical study within 6 weeks prior to study start
* have participated in another Baxter vaccine study in the past 6 months (with the exception of follow-up studies)
* For female subjects: pregnancy or lactation

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-05; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Principal Investigator — Baxter BioScience
Locations (1):
- SGS Biopharma Research Unit Stuivenberg, Antwerp, Belgium

REFERENCES:
- [Derived] Orlinger KK, Hofmeister Y, Fritz R, Holzer GW, Falkner FG, Unger B, Loew-Baselli A, Poellabauer EM, Ehrlich HJ, Barrett PN, Kreil TR. A tick-borne encephalitis virus vaccine based on the European prototype strain induces broadly reactive cross-neutralizing antibodies in humans. J Infect Dis. 2011 Jun 1;203(11):1556-64. doi: 10.1093/infdis/jir122. PMID 21592984